CLINICAL TRIAL: NCT02486913
Title: Enhancing the Diagnosis and Prevention of Cardiovascular Disease in Newham by Integrated Use of Electronic Health Records
Brief Title: Enhancing Diagnosis and Prevention of Cardiovascular Disease in Newham by Integrated Use of Electronic Health Records
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MCPH1C8R
Record Dates: First submitted 2015-06-16; First posted 2015-07-01 (Estimated); Last update posted 2018-03-06 (Actual); Status verified 2017-02

CONDITIONS: Cardiovascular Disease
Keywords: Primary prevention; National Health Service Health Check
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional Health Check (No Intervention): Patients undergoing conventional National Health Service Health Check
- Enhanced Health Check (Experimental): Patients undergoing National Health Service Health Check enhanced by risk report
  Interventions: Other: Enhanced Health Check

INTERVENTIONS:
Other: Enhanced Health Check — National Health Service Health Check enhanced by risk report
  Arms: Enhanced Health Check

SUMMARY:
The investigators will develop a "risk report" within the primary care electronic health record (EMIS) for patients attending for their National Health Service Health Check. The value of the report for reducing cardiovascular risk will be assessed qualitatively and also quantitatively in a non-randomised comparative trial.

DETAILED DESCRIPTION:
The investigators will design a template within the primary care electronic health record (EMIS) that draws on Health Check data to provide a contemporary "risk report". Included in the report will be clear description of life-time cardiovascular risks, the factors driving those risks and how risk might be reduced through life-style and risk factor modification. The investigators will evaluate the benefits of providing patients with a risk report qualitatively by patient and clinician interviews. Quantitative analysis of the benefit of the risk report will be provided by a non-randomised comparative trial. First, a group of patients undergoing a conventional Health Check will be recalled after three months for a second Health Check, allowing measurement of the change in "Heart Age" - a convenient index of life-time cardiovascular risk. Following introduction of the risk report the investigators will recall a further group of patients for a second Health Check, allowing measurement of the change in "Heart Age". The effect of the risk report will be determined by comparing the change in Heart Age between the two groups of patients.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 40-74 years

Exclusion Criteria:

* Prior diagnosis of heart disease, stroke, diabetes, kidney disease or dementia

Ages: 40 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2015-08; Primary Completion 2018-01-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Change in Heart Age | 3 months
  Change in Heart Age between 1st Health Check and 2nd Health Check three months later

SECONDARY OUTCOMES:
Changes in smoking status | 3 months
  Changes in smoking status (number smoked per day) by direct patient enquiry between 1st Health Check and 2nd Health Check three months later.
Change in total cholesterol | 3 months
  Changes in total blood cholesterol (mmol/L) by serum sampling between 1st Health Check and 2nd Health Check three months later.
Change in systolic blood pressure | 3 months
  Change in systolic blood pressure (mmHg) by direct measurement using an inflatable cuff between 1st Health Check and 2nd Health Check three months later.
Change in body mass index | 3 months
  Change in body mass index by measurement of height and weight between 1st Health Check and 2nd Health Check three months later.

CONTACTS AND LOCATIONS:
Overall Officials: Adam D Timmis, MD FRCP, Principal Investigator — Queen Mary University of London
Locations (1):
- Bart's Heart Centre, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hawking MKD, Timmis A, Wilkins F, Potter JL, Robson J. Improving cardiovascular disease risk communication in NHS Health Checks: a qualitative study. BMJ Open. 2019 Sep 3;9(8):e026058. doi: 10.1136/bmjopen-2018-026058. PMID 31481364
- See also: NHS Health Check Home Page — http://www.healthcheck.nhs.uk/